CLINICAL TRIAL: NCT02093936
Title: Lymphocytes Cut Off Values of Induced Sputum Samples in Healthy and Non-healthy Patients- A Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-14-SK-0629-13-CTIL
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Respiratory Tract Diseases; Occupational Diseases; Disorders of Environmental Origin
Keywords: airway inflammation; induced sputum; normal values; lymphocyte; eosinophil; neutrophil
MeSH Terms: conditions — Respiratory Tract Diseases; Occupational Diseases; Disorders of Environmental Origin

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy non exposed: Healthy patients with no pulmonary symptoms that were not exposed to occupational or environmental exposure
- Healthy exposed: Healthy patients with no pulmonary symptoms that were exposed to occupational or environmental exposure
- Non-healthy exposed: Patients with pulmonary symptoms or diseases that were exposed to occupational or environmental exposure
- Non-healthy non-exposed: Patients with pulmonary symptoms or diseases that were not exposed to occupational or environmental exposure

SUMMARY:
Background: Induced sputum (IS) is a noninvasive methodology for evaluating airway inflammation in a large number of pulmonary diseases, i.e, Asthma, Chronic obstructive pulmonary disease and Interstitial Lung Diseases. Several studies have defined normal values and cut-off points for this technique based on cellular components of IS, such as percentages of eosinophils, neutrophils, macrophages and CD4/CD8 ratio of T cell lymphocytes. However, normal values and cut-off points for lymphocyte percentages indicative of pathology have not yet been established or validated. This component of IS has considerable clinical value. Similar to other constituents of IS, it can provide biological insights into the pathogenesis of respiratory disorders and contribute to establishing the diagnosis and guiding treatment management of a variety of airway diseases.

The purposes of this study are to define normal values and cut-off points of lymphocytes in IS among individuals with respiratory disorders and healthy volunteers, and to verify the current reference values of the percentage of eosinophils, neutrophils and CD4/CD8 ratio in IS.

Methods: A Cross Sectional study which includes a database on up to 900 patients who participated in various studies conducted in the Pulmonary Laboratory of Tel Aviv Sourasky Medical Center between 2005 to 2012 will be established. The study population will include patients diagnosed as having various pulmonary diseases and a group of healthy volunteers who will serve as controls. The cut-off for normal values of lymphocyte, eosinophil and neutrophil percentages and CD4/CD8 ratio in IS will be defined by using ROC curves and evaluating sensitivity and specificity. The comparison of the different values to those in the literature will be done by using the Spearman rank correlation.

The results of this study will provide supplementary information on lymphocyte counts in IS for identifying and treating various respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from pulmonary symptoms or diseases
* patients with occupational or environmental exposure

Exclusion Criteria:

* indefinite spirometry tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who were sent to the Pulmonology and Allergy Laboratory in the Tel Aviv sourasky medical center between the years 2005-2012. Some had a certain occupational or environmental exposue, some had pulmunary symptoms or diseases and some had both of the above. They were sent in order to examine through spirometry and induced sputum tests wheather they suffer from a pulmonary pathology.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-01; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Healthy patients vs. non-healthy patients | 1 year
  Healthy patients are those who did not suffer from major respiratory symptoms, were not diagnosed with any pulmonary diseases and had normal pulmonary function tests (i.e, FEV1>80%, FEV1/FVC ratio>75%).
  Non-healthy patients are those who suffered from respiratory symptoms, were diagnosed with a pulmonary disease or had abnormal pulmonary function tests (i.e, FEV1<80%, FEV1/FVC ratio<75%).

SECONDARY OUTCOMES:
Eosinophil percentage out of all White blood cells in Sputum sample | Up to 1 day from sputum induction
Neutrophil percentage out of all White blood cells in Sputum sample | Up to 1 day from sputum induction
T cell Lymphocyte cluster of differentiation 4 / cluster of differentiation 8 (CD4/CD8) ratio in Sputum sample | Up to 1 day from sputum induction
Lymphocyte percentage out of all White blood cells in Sputum sample | Up to 1 day from sputum induction

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Kivity, Professor, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel, Israel

REFERENCES:
- [Background] Balbi B, Pignatti P, Corradi M, Baiardi P, Bianchi L, Brunetti G, Radaeli A, Moscato G, Mutti A, Spanevello A, Malerba M. Bronchoalveolar lavage, sputum and exhaled clinically relevant inflammatory markers: values in healthy adults. Eur Respir J. 2007 Oct;30(4):769-81. doi: 10.1183/09031936.00112306. PMID 17906085
- [Background] Fireman Z, Osipov A, Kivity S, Kopelman Y, Sternberg A, Lazarov E, Fireman E. The use of induced sputum in the assessment of pulmonary involvement in Crohn's disease. Am J Gastroenterol. 2000 Mar;95(3):730-4. doi: 10.1111/j.1572-0241.2000.01843.x. PMID 10710066
- [Background] Fireman E, Topilsky I, Greif J, Lerman Y, Schwarz Y, Man A, Topilsky M. Induced sputum compared to bronchoalveolar lavage for evaluating patients with sarcoidosis and non-granulomatous interstitial lung disease. Respir Med. 1999 Nov;93(11):827-34. doi: 10.1016/s0954-6111(99)90269-x. PMID 10603633
- [Background] Fireman E, Boikaner T, Priel IE. Combined CD4/CD8 ratio in induced sputum and pulmonary function testing for non-invasive identification of sarcoidosis. Transl Res. 2006 Aug;148(2):87-95. doi: 10.1016/j.trsl.2006.03.005. PMID 16890149
- [Background] Pin I, Gibson PG, Kolendowicz R, Girgis-Gabardo A, Denburg JA, Hargreave FE, Dolovich J. Use of induced sputum cell counts to investigate airway inflammation in asthma. Thorax. 1992 Jan;47(1):25-9. doi: 10.1136/thx.47.1.25. PMID 1539140